CLINICAL TRIAL: NCT07325994
Title: Verbal Analgesia Versus Standard Care for Pain Control in Women With Primary Infertility Undergoing Vaginoscopic Office Hysteroscopy: A Randomized Controlled Trial
Brief Title: Verbal Analgesia Versus Standard Care for Pain Control in Women With Primary Infertility Undergoing Office Hysteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, Clinical Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: verbal analgesia Hysteroscopy
Record Dates: First submitted 2025-09-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal analgesia (Experimental): Providers will deliver a standardized verbal analgesia script in a calm, slow-paced, supportive tone, synchronized to procedural steps:
  * Scope introduction (introitus → external os): "You may feel light pressure as the camera enters-keep a slow, steady breath; you are doing well."
  * Cervical passage (internal os): "A brief pinch or cramp may happen now; it will pass quickly-breathe in slowly, and out."
  * Uterine entry and distension: "A feeling of fullness is expected; stay with your breath-it eases in moments."
  * Cavity inspection: "You may notice short waves of cramp; they are normal and brief-you're managing this well."
  * Withdrawal: "We are nearly finished-slow exhale as we come out. That's it, you did great." Providers will undergo training to ensure fidelity. All participants will receive ibuprofen 600 mg orally one hour before hysteroscopy as standard analgesia.
  Interventions: Behavioral: verbal analgesia
- standard care (Sham Comparator): Providers will use neutral, procedural statements without supportive phrasing, e.g., "Starting the camera now," "Passing the cervix," "Entering the uterus," "Inspecting the cavity," "Withdrawing the camera." All participants will receive ibuprofen 600 mg orally one hour before hysteroscopy as standard analgesia.
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: verbal analgesia — Providers will deliver a standardized verbal analgesia script in a calm, slow-paced, supportive tone, synchronized to procedural steps:
  * Scope introduction (introitus → external os): "You may feel light pressure as the camera enters-keep a slow, steady breath; you are doing well."
  * Cervical passage (internal os): "A brief pinch or cramp may happen now; it will pass quickly-breathe in slowly, and out."
  * Uterine entry and distension: "A feeling of fullness is expected; stay with your breath-it eases in moments."
  * Cavity inspection: "You may notice short waves of cramp; they are normal and brief-you're managing this well."
  * Withdrawal: "We are nearly finished-slow exhale as we come out. That's it, you did great." Providers will undergo training to ensure fidelity. All participants will receive ibuprofen 600 mg orally one hour before hysteroscopy as standard analgesia.
  Arms: Verbal analgesia
Behavioral: standard care — Providers will use neutral, procedural statements without supportive phrasing, e.g., "Starting the camera now," "Passing the cervix," "Entering the uterus," "Inspecting the cavity," "Withdrawing the camera.". All participants will receive ibuprofen 600 mg orally one hour before hysteroscopy as standard analgesia.
  Arms: standard care

SUMMARY:
Office hysteroscopy is a cornerstone in the diagnostic evaluation of infertile women, enabling direct visualization of the uterine cavity for identifying intrauterine pathology. The vaginoscopic ("no-touch") approach, which eliminates the use of a speculum and tenaculum, is increasingly adopted due to improved tolerability, higher success rates, and reduced pain compared to conventional methods.

DETAILED DESCRIPTION:
Office hysteroscopy is a cornerstone in the diagnostic evaluation of infertile women, enabling direct visualization of the uterine cavity for identifying intrauterine pathology. The vaginoscopic ("no-touch") approach, which eliminates the use of a speculum and tenaculum, is increasingly adopted due to improved tolerability, higher success rates, and reduced pain compared to conventional methods.

Despite this, many women still report moderate to severe pain, particularly during cervical passage and uterine distension. High pain scores may result in incomplete examinations, decreased patient satisfaction, and increased need for sedation or analgesia. Various pharmacological interventions have been studied, including NSAIDs, local anesthetics, and misoprostol, with inconsistent or limited benefit.

Verbal analgesia, a structured communication strategy involving calm, supportive, and reassuring verbal cues, has been shown to reduce procedural pain in other gynecologic settings such as IUD insertion. However, no randomized trial has specifically evaluated structured verbal analgesia in women with primary infertility undergoing vaginoscopic office hysteroscopy. This trial aims to address this evidence gap by comparing verbal analgesia with standard neutral communication, with both groups receiving baseline NSAID premedication.

ELIGIBILITY:
Inclusion Criteria:

* o Women aged 18-40 years.

  * Diagnosis of primary infertility (failure to conceive after ≥12 months of unprotected intercourse).
  * Indication for diagnostic office hysteroscopy.
  * Regular menstrual cycles.

Exclusion Criteria:

* o Secondary infertility.

  * Known pelvic infection, cervicitis, or vaginitis.
  * Use of analgesics within 8 hours prior to procedure.
  * Cervical stenosis, prior failed hysteroscopy, or known uterine anomaly.
  * Contraindication to NSAIDs
  * Pregnancy or suspected pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
pain during OH | During the procedure (immediately after insertion of hysteroscope, assessed within 5 minutes
  It will be measured by 0-10 numerical rating scale where 0 indicates no pain and 10 worst pain imaginable

SECONDARY OUTCOMES:
Patient satisfaction | At the end of the visit (within 30 minutes of procedure completion)
  Patient satisfaction on a 0-10 NRS (0 = no satisfaction, 10 = maximum satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Al Gezeera Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided